CLINICAL TRIAL: NCT03906162
Title: A 12-week Intervention With Motivational Interviewing and Physical Activity Monitoring, to Enhance the Daily Amount of Physical Activity in Community Dwelling Older Adults - a Randomized Controlled Trial
Acronym: MIPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Rasmus Tolstrup Larsen, Principal investigator, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18004960
Record Dates: First submitted 2019-04-01; First posted 2019-04-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Aging; Physical Activity; Older Adults
Keywords: physical activity monitors; motivational interviewing; walking; fitness-tracker; social cognitive theory; older age
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 12 week intervention with two groups in a parallel design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Primary investigator will be blinded for allocation before making the final analyses. No outcome assessments will be made by an assessor. Only objectively measured steps per day and participant reported outcome measures will be used for this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental): Experimental content + base intervention
  Interventions: Behavioral: Motivational interviews; Behavioral: Base intervention
- Control intervention (Active Comparator): Base intervention
  Interventions: Behavioral: Base intervention

INTERVENTIONS:
Behavioral: Motivational interviews — During the 12-week intervention, the participants will receive seven telephone calls from a physical therapist. The interviews will be held in week 1, 2,3,5,7,9, and 12.
  The telephone call will consist of a motivational interview focused on enhancing the daily level of physical activity in the participants.
  MI is a form of counselling aiming at prompting increases in self-efficacy, which may leave people more open to and invested in changing their behaviours and shows potential for significant effects for exercise behaviour change.
  In addition to the telephone based motivational interviews, the experimental group will also receive the "base intervention" which is described in detail under the "control intervention paragraph".
  Arms: Motivational interviewing
Behavioral: Base intervention — The "base intervention" consists of a physical activity monitor (PAM) for everyday use in the intervention period and a pamphlet with information about Danish recommendations on physical activity in aging populations. The PAM will be the Garmin Vivofit 3 monitor linked to a pre-specified Garmin Connect account. The participants will be asked to install the Garmin Connect application on their smartphone and use the given ID/password in the app. The participants will be asked to wear the monitor 24-hours a day for the 12-week intervention period. The participants can use the PAM as they like but they will be asked to try to use the PAM and the application to enhance their daily level of physical activity.

SUMMARY:
To investigate if motivational-interviewing will enhance the expected effect from physical activity monitors, on physical activity in older adults, we will conduct a two-arm randomized controlled trial in 2019.

Both groups in the trial will receive a physical activity monitor for everyday use in the 12-week intervention period and a folder with information about the benefits of physical activity in older age. Participants in the intervention group will in addition to the use of the physical activity monitors receive a motivational feedback session by phone of about 20 minutes constructed from the theoretical framework of Motivational interviewing by Rollnick, Miller & Butler and Social Cognitive Theory by Bandura. The content of the session focuses on investigating the most relevant possibilities and barriers for the participant to increase his or her levels of PA.

The primary outcome will be between group difference in average steps per day throughout the intervention period, measured objectively by the physical activity monitor (Garmin Vivofit 3). Secondary outcomes include participant reported outcome measures such as 'International Physical Activity Questionnaire', 'Nordic Physical Activity Questionnaire', 'EQ5D Quality of life questionnaire', 'UCLA Loneliness Scale', 'Self Efficacy for Exercise', and 'Outcome expectancy for Exercise'. To ensure 80% power with an alpha-level on 0.05, we will include 128 participants. The study will enroll in March 2019.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Be minimum 70 years of age at the time of inclusion
* Own and use an Apple/Google/Microsoft smartphone device compatible with the Garmin Connect™ Mobile application.
* Own use an e-mail account
* Live in Denmark and have a Danish postal address and be able to receive the intervention content.
* Be able to walk independently with or without assistive devices.

Exclusion Criteria:

Participants cannot

* Receive active cancer treatment
* Have major cognitive impairment (e.g. dementia or alzheimers).
* Parkinson's or Multiple Sclerosis (or similar disease) affecting their mobility in such a way that the participants cannot walk on a daily basis.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Individual intervention period average of PAM measured steps per day | A daily average of the 12 weeks of intervention
  Daily step counts will be objectively measured by the PAM.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Baseline + end point at 12 weeks + follow up at 6 months and 12 months
  Questionnaire: The seven-item IPAQ-SF measure assesses the types of intensity of physical activity and sitting time that people has done the past seven days as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
Nordic Physical Activity Questionnaire | Baseline + end point at 12 weeks + follow up at 6 months and 12 months
  Questionnaire: It is developed to monitor compliance with the WHO recommendations on PA.
EQ5D Quality of life questionnaire | Baseline + end point at 12 weeks + follow up at 6 months and 12 months
  Questionnaire: The EQ-5D-5L is a generic health-related quality of life (HRQoL) measure developed as a non-disease-specific instrument for describing and valuing health states and comprises five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each of which has three levels (no problems, moderate problems and extreme problems) and a visual analogue scale (EQ VAS). The score for the five dimensions can be combined into a five-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
University of California, Los Angeles, Loneliness Scale | Baseline + end point at 12 weeks + follow up at 6 months and 12 months
  Questionnaire: The 20-item UCLA loneliness scale (third version) is a self-report measure of loneliness and social isolation. The scale consists of 11 positive and nine negative items and the total score is calculated by finding the sum of 20 items (0-60), with a higher score indicating more loneliness.
Self Efficacy for Exercise | Baseline + end point at 12 weeks + follow up at 6 months and 12 months
  Questionnaire: The nine-item SEE-DK addresses confidence to engage in regular exercise [44], when challenged by known barriers to exercise. The scale was developed initially for sedentary adults in the community who participated in an outpatient exercise program and was revised to older adults. It is designed to be administered using face-to-face interview. Response categories range from 0 (no confidence) to 10 (very confident). Item scores are used to calculate a total score (0-90), with higher scores indicating higher confidence, or self-efficacy, related to exercise. The SEE-DK is adapted to Danish older adults with acceptable face and content validity, construct validity by acceptable model fit as a unidimensional scale, and test-retest reliability.
Outcome expectancy for Exercise | Baseline + end point at 12 weeks + follow up at 6 months and 12 months
  Questionnaire: The 13-item OEE-2 scale was developed from the original 9-item Outcome Expectations for Exercise scale (OEE) that specifically focused on measuring the positive outcome expectations for exercise (POEE). To complete the OEE2-DK scale the participants are asked, using a Likert scale, to strongly agree, agree, neither agree nor disagree, disagree, or strongly disagree with the stated outcomes to each statement of exercising.

CONTACTS AND LOCATIONS:
Locations (1):
- Rasmus Tolstrup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised data set will be published with the published paper
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Five years from published paper

REFERENCES:
- [Derived] Larsen RT, Korfitsen CB, Keller C, Christensen J, Andersen HB, Juhl C, Langberg H. The MIPAM trial - motivational interviewing and physical activity monitoring to enhance the daily level of physical activity among older adults - a randomized controlled trial. Eur Rev Aging Phys Act. 2021 Jul 2;18(1):12. doi: 10.1186/s11556-021-00269-7. PMID 34215176
- [Derived] Larsen RT, Korfitsen CB, Juhl CB, Andersen HB, Christensen J, Langberg H. The MIPAM trial: a 12-week intervention with motivational interviewing and physical activity monitoring to enhance the daily amount of physical activity in community-dwelling older adults - a study protocol for a randomized controlled trial. BMC Geriatr. 2020 Oct 20;20(1):412. doi: 10.1186/s12877-020-01815-1. PMID 33081715

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT03906162/Prot_SAP_ICF_001.pdf